CLINICAL TRIAL: NCT04496635
Title: Evaluation of the Application and Efficacy of Prevention Measures for Surgical Site Infection in Elective Colorectal Surgery.
Brief Title: Surveillance and Implementation of a Bundle of Care to Reduce Surgical Site Infection in Colorectal Surgery (CCR-VINCat)
Acronym: CCR-VINCat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Granollers (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CCR-VINCat 1
Record Dates: First submitted 2020-07-14; First posted 2020-08-03 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Colon Rectal Cancer; Surgical Site Infection
Keywords: Surveillance; Preventative measures; Bundle of care; Colorectal surgery; Surgical site infection; Prevention
MeSH Terms: conditions — Colonic Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: The study compare two phases: baseline (BP), from 2008 to 2015, and implementation (IP), from 2016 to 2018.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline phase (No Intervention): Patients included in the VINCat program, and operated on colorectal surgery between 2007 and 2015 in Catalonia
- Implementation phase (Experimental): Patients included in the VINCat program, and operated on colorectal surgery between 2016 and 2018 in Catalonia
  Interventions: Other: Implementation of a bundle of care

INTERVENTIONS:
Other: Implementation of a bundle of care
  Arms: Implementation phase

SUMMARY:
The Nosocomial Infection Surveillance Program in Catalonia (VINCat) monitors surgical site infection (SSI) in elective colorectal surgery since 2007 in 55 public and private acute care hospitals. These hospitals perform active and prospective standardized surveillance of elective colorectal resections. Post-discharge surveillance is mandatory at least up to 30 days after surgery. Hospitals are classified according to their size into three groups: >500 hospital beds; 200-500 beds; <200 beds.

Aim. To examine the effect on SSI rate of a specific preventative bundle in elective colorectal surgery.

Methods. Pragmatic study using VINCat prospective colorectal database from 2007 to 2018. In 2016, a bundle of six preventative measures was recommended to the VINCat hospitals.

To compare the results of SSI before (baseline phase, BP) and after the bundle implementation (implementation phase, IP) a logistic regression model has been established. The results will be shown as Odds Ratio (OR) and the corresponding confidence intervalsCI95. The significance level will be fixed at 5% (P < 0.05).

DETAILED DESCRIPTION:
Surveillance. The VINCat Program was developed in the 2007 as the Nosocomial Infection Surveillance system in Catalonia, covering a population of seven and a half million people. The system is similar to other international reference programs, such as the National Healthcare Safety Network (NHSN), and its described in detail on the VINCat website. Hospitals carry out active and prospective standardized surveillance, and are classified according to their number of beds into three groups: group 1 (500 beds); group 2 (200-500 beds); group 3 (200 beds). The staff performing surveillance had received training in the VINCat surveillance methodology to ensure the collection of homogeneous, accurate data.

Surveillance is continued at least for 30 days after the operation. All public and private participating hospitals report data voluntarily and receive feedback once a year.

Monitoring of colorectal surgery is performed prospectively and continued until a minimum of 100 interventions per year is reached in each hospital, although some centres include all their yearly cases. Hospitals with less than 10 interventions per year are excluded. Participating hospitals record the data on an Internet-based database.

Follow-up and post-discharge surveillance. Patients are followed up by trained infection control staff. Active mandatory post-discharge surveillance is performed at least to day 30 post surgery by a multimodal approach including electronic review of clinical records (primary and secondary care), checking readmissions, checking emergency visits, and reviewing microbiological and radiological data.

Development of the colorectal surgical site infection program. In 2015, a multidisciplinary team of nurses and medical specialists from the VINCat Program, and surgeons belonging to the Catalan Society of Surgery was set up to formulate a specific bundle of SSI preventative measures for colorectal surgery. The literature for optimal care during the preoperative, intraoperative and postoperative phases was reviewed, including evidence on oral antibiotic prophylaxis and mechanical bowel preparation. Practices were chosen either by their high levels of scientific evidence or by being considered, by consensus, reasonable, associated with minimal risk, and potentially beneficial.

The working group developed a 6 measures bundle to be voluntary implemented by the participating hospitals. The measures of the bundle are: intravenous and oral antibiotic prophylaxis, mechanical bowel preparation (MBP), laparoscopic surgery, maintenance of normothermia, and the use of a wound retractor.

The intervention began on 1 January 2016, with diffusion of the bundle measures via e-mail, and a workshop addressed to all to the surgical and ICT teams.

Definitions. SSI is defined according to the Centers for Disease Control (CDC) and is stratified into categories of surgical procedures (-1 to 3) according to the risk of surgical infection defined by the NHSN.

Design of the pragmatic trial. Implementation of the bundle precluded randomization. The study compared two phases: baseline (BP), from 2008 to 2015, and implementation (IP), from 2016 to 2018.

Fifty-five of the 66 hospitals participating in the VINCat Program were included in the analysis. Prospective surveillance was performed by the infection control team (ICT) of each hospital to ensure appropriate data collection. The surveillance period lasted from January 2007 to December 2018. During the first 4 years of the program, the results of colon and rectal surgery were aggregated. From 2011, data is separated for each type of surgery.

As all eligible patients were included in the pragmatic design, informed consent was not obtained.

The study was conducted as a performance improvement project and approved by the Ethics in Research Committee.

Statistical analysis Data will be summarized as frequencies and proportions for categorical variables or as medians and interquartile range (IQR) for continuous variables. Infection rates will be expressed as cumulative incidence, that is, the crude percentage of operations resulting in SSI/ number of surgery procedures. Data will be also stratified by year, risk index category, hospital group and SSI type.

To analyse the relationship between two qualitative variables, contingency tables will be used, and the chi-square test or the likelihood ratio test will be performed. The analysis will be completed with grouped bar graphs. To analyse differences in the proportion of infection over the years, the logistic regression model will be performed. The results will be presented in terms of OR or estimated infection rates, with the corresponding 95% confidence intervals. The significance level will be set at 5% in all tests. The results will be analysed using software: Statistical Analysis Systems (SAS) v9.4, SAS Institute Inc., Cary, USA.

ELIGIBILITY:
Inclusion Criteria:

* Colon or rectal elective surgery.

Exclusion Criteria:

* Peritonitis at the time of intervention ("dirty" surgery) Patients who underwent multiple procedures during the same surgery, for example resection of liver metastases Centers that performed less tan 10 surgical procedures annually Centers that have not been able to ensure prospective surveillance during hospitalization or effective monitoring of cases within 30 days of the intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60000 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection rate | 30 days
  Overall surgical infection rate

SECONDARY OUTCOMES:
Organ/space surgical infection rate | 30 days
  Specific organ/space surgical infection rate
Hospital type-Surgical infection rate | 30 days
  Comparison of rates among the three hospitals groups, according to their size
Analysis (logistic regression model) of the efficacy of each preventive measure | 30 days
  Univariate and multivariate logistic regression to analise the efficacy of each individual measure belonging to the bundle of care.

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Badia-Perez, MD, PhD, Principal Investigator — Fundació Hospital General de Granollers
Locations (1):
- Hospital General de Granollers, Granollers, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be shared when requested